CLINICAL TRIAL: NCT06465823
Title: A Phase 2 Double Blind Placebo Controlled Study on the Efficacy of Bumetanide for Cognitive Improvement in Children and Adolescents With Down Syndrome
Brief Title: Efficacy of Bumetanide to Improve Cognitive Functions in Down Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stefano Vicari (Other)
Collaborators: Italian Institute of Technology (IIT) (Unknown)
Responsible Party: Sponsor-Investigator, Stefano Vicari, Stefano Vicari - Head of Child and Adolescent Neuropsychiatry Unit, Bambino Gesù Hospital and Research Institute
Organization: Bambino Gesù Hospital and Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1042_OPBG_2016
Record Dates: First submitted 2024-05-06; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Down Syndrome
Keywords: Bumetanide, GABA, NKCC1, Memory
MeSH Terms: conditions — Down Syndrome | interventions — Bumetanide

STUDY DESIGN:
Intervention Model Description: This is a double-blind placebo-controlled study. The enrolment will include 64 patients. Children and adolescents with DS (aged 10-17) will be assigned to one of the two conditions by an automated process: Bumetanide treatment or control group, by a stratified random sampling based on the mental age (≥ 4.5 age <5.5 yrs vs ≥5.5 age < 8.5yrs). Patients in the Bumetanide group will be treated for 3 months with a dose of 0.02 mg/kg twice a day, oral administration. Patients in the control group will be administered a placebo. The randomization will be conducted during the first appointment after the informed consent has been signed, and the inclusion and exclusion criteria have been verified.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The responsible for the collection of the assessments or evaluator will remain blind to treatment allocation during the trial and primary analyses. The diuretic actions of Bumetanide may impact the blinding procedure. To reduce this impact, the psychologist evaluator will be separated from the pediatrician who will treat the children, thus ensuring the blindness to the treatment. A supervisor during each assessment session will control for any possible interference with the evaluator's blindness. The randomization schedule will be kept inaccessible to the personnel involved in the study. In cases of serious adverse effects, the envelope will only be opened by the Principal Investigator who will be the only one to know the treatment assignment. The Principal Investigator will ensure that the contents of the envelope are kept in a place inaccessible to others.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bumetanide (Experimental): Patients in the experimental group will receive the pharmacological treatment with Bumetanide
  Interventions: Drug: Bumetanide
- Placebo (Placebo Comparator): Patients in the control group will receive the placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bumetanide — Patients in the Bumetanide group will be treated for 3 months with a dose of 0.02 mg/kg twice a day, oral administration. It will be labeled (pre-printed and indistinguishable) with the randomization number and site number and will be delivered in separate blocks during the first, second and fourth appointment.
  The patients will start the treatment with half of the full target dose during the first week:
  * If the target dose is 0.5mg BID, only the morning dose will be administrated.
  * If the target dose is 1.0 mg BID the dose will be 0.5 mg BID.
  * If the target dose is 1.5mg BID, the morning dose will be 1.0 mg, the evening dose will be 0.5 mg.
  * If the target dose is 2.0 mg BID the dose will be 1.0 mg BID The patient will continue with the full dose starting from Visit 2 after 1 week of dosing.
  Arms: Bumetanide
Drug: Placebo — Patients in the control (placebo) group will be given placebo for 3 months twice a day, oral administration. The Placebo tablets will be visually indistinguishable from Bumetanide and packaged as Bumetanide. The placebo will be labeled (pre-printed and indistinguishable) with the randomisation number and site number and will be delivered in separate blocks during the first, second and fourth visits.
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the clinical efficacy of a known diuretic drug, Bumetanide, in terms of improvement of memory and psychological functioning in children and adolescents with Down syndrome (DS), in order to develop therapeutic strategies for cognitive and psychopathology aspects associated with the syndrome. The study also aims to identify possible predictors and biological and genetic markers related to the efficacy of the treatment. Recently, preliminary studies conducted on the animal model of Down syndrome have proven the efficacy of the drug Bumetanide in counteracting some brain anomalies related to communication between nerve cells (synaptic transmission) typical of the syndrome, with the effect of improving memory skills. Behaviour-enhancing effects have also been found in preliminary studies in humans with other neurodevelopmental disorders (e.g., autism spectrum disorders). The drug Bumetanide could therefore be useful in counteracting the biological mechanisms that cause some cognitive deficits associated with Down syndrome. The potential of this therapeutic approach will be tested through a clinical trial in a population of children and adolescent patients with DS, in a randomized placebo-controlled trial with a three-month treatment with Bumetanide. Participants will be randomly assigned to the experimental group that will receive the treatment (Bumetanide) vs the control/comparison group that will receive the placebo. Bumetanide is a diuretic drug that has been widely used in humans in the past with few side effects, is orally active, and is very inexpensive. 64 participants will be recruited.

DETAILED DESCRIPTION:
Down syndrome (DS) is a leading cause of genetically defined intellectual disability. It is characterized by low IQ and cognitive deficits, especially learning and memory. Among the neurobiological causes of these deficits, the increased generation of GABAergic interneurons in the forebrain during development is thought to impair learning and memory in Ts65Dn mice, inducing excessive inhibition and a consequent imbalance of excitatory/inhibitory signals. This derangement would affect cognition in Ts65Dn mice by altering hippocampal synaptic plasticity. Indeed, both LTP and cognitive deficits can be improved by reducing the GABA-mediated signal strength through GABAAR antagonist treatment. Some studies on animal models have helped to demonstrate that the use of an inhibitor of the NKCC1 pump such as Bumetanide helps to restore the imbalance of the GABAergic signal and the synaptic plasticity of the hippocampus with a consequent improvement in memory and learning abilities even after only one treatment week. Recently, the modulation of the GABAergic signal by inhibiting the activity of the NKCC1 pump, a specific inhibitor such as Bumetanide, has demonstrated enormous potential for improving epileptic symptoms and autistic symptoms (disorders associated with an imbalance of the excitatory/inhibitory synaptic signal) in animal models and humans and of memory deficits in DS animal models. The hypothesis of the study is therefore that the use of Bumetanide can counteract the alterations of the cerebral GABAergic signal in people with DS, improving their cognitive and psychological abilities. This is a non-profit phase II randomized placebo-controlled study involving 64 participants. The study for each patient will be concluded at the end of treatment (at 3 months) and follow-up (at 5 months). In general, the study will be concluded with the follow-up visit of the last 64th patient. The enrollment of patients will last one year and will take place, like all the visits foreseen by the trial, only at the IRCCS Bambino Gesù Pediatric Hospital in Rome - Trials Complex Operative Unit. For some biomarker analyses, the study makes use of collaboration with the Italian Institute of Technology and the Giannina Gaslini Institute of Genoa. Participation in the study includes an initial visit to verify that the subject's condition meets the criteria required by the study. Subsequently, six follow-up visits will be scheduled after 1 week, 2 weeks, 1 month, 2 months, 3 months (end of treatment), and 2 months after the end of treatment (after 5 months from the start of treatment). Bumetanide drug and placebo (indistinguishable) will be dispensed to participants during the first (Day 1), second (Day 7± 1), and fourth visit (Day 31± 3). Participants in the Bumetanide group will be treated for three months with a dose of 0.02 mg/kg twice a day orally. Participants in the control group will take a placebo twice a day for three months orally. All participants in the study will undergo instrumental and laboratory tests according to the schedule and times indicated below:

* Psychological and neuropsychological evaluation at the time of recruitment (at the first visit - Day 1), at the end of treatment (after three months - Day 31± 3), and two months after the end of treatment (after five months from the start of treatment - Day 150 ± 4). This evaluation will be carried out through long-term memory tasks, executive functions measures and adaptive level, and through scales and interviews on the psychopathological aspects and will be important for evaluating the effects of the treatment. The first visit includes cognitive level assessment (Day 1).
* Questionnaire on quality of life, sleep, and stool and the analysis of vital signs will be performed at the first visit on Day 1, after one week (Day 7± 1), after one month (Day 31± 3), after three months (Day 90 ± 3) and after two months from the conclusion (five months from the start of treatment - (Day 150 ± 4).
* Physical examination in the first visit (Day 1), after one week (Day 7± 1), after one month (Day 31± 3), after three months (Day 90 ± 3), after two months from the conclusion of the treatment (five months from the beginning of the treatment- Day 150 ± 4).
* Blood sampling, specifically, for the analysis of electrolytes and blood gas and for hemogenic and liver function tests during all visits (Day 1 Day 7± 1, Day 15± 1, Day 31± 3, Day 61± 3, Day 90 ± 3, Day 150 ± 4 ). •Urine analysis at first visit (Day 1 during all visits (Day 1 Day 7± 1, Day 15± 1, Day 31± 3, Day 61± 3, Day 90 ± 3, Day 150 ± 4).
* Audiometric test at the start of treatment (Day 1), after one month (Day 31± 3), after three months (end of treatment - Day 90 ± 3) and two months after the end of treatment (five months after start of treatment - Day 150 ± 4). • Electrocardiogram (ECG) at the first visit (Day 1), after one week (Day 7± 1), after one month (Day 31± 3), after three months (end of treatment - Day 90 ± 3), and two months after the end of treatment (five months after starting treatment - Day 150 ± 4).
* Electroencephalogram (EEG) at the first visit (Day 1), after one month (Day 31± 3) after three months (end of treatment - Day 90 ± 3), and two months after the end of treatment (five months after the start of treatment - Day 150 ± 4).
* Nephrological evaluation at first visit (Day 1), after one week (Day 7± 1), after two weeks (Day 15± 1), after one month (Day 31± 3), after two months and at the end of treatment (after three months - Day 90 ± 3).
* Pregnancy test for girls before starting treatment (Day-1).

The study also predict safety measures. Adverse events will be recorded using the UKU side effect rating scale. Furthermore, participants will be closely monitored by Investigators during critical periods before, during and after the treatment.

ELIGIBILITY:
Principal inclusion criteria

1. The presence of a free trisomy 21 documented by karyotyping
2. Adolescents from 10 to 17 years old (included)
3. 3 4.5 ≥ Mental age ≤ 8.5 (as assessed by Leiter-3 at visit 1 or by assessment with Leiter-3 within 6 months of the first visit (Visit 1)
4. Informed consent from their parents and assent from child/adolescent

Principal exclusion criteria

1. The presence of any neurosensory deficits, such as hypoacusis or serious visual impairments;
2. The presence of epilepsy;
3. The presence of electrolyte disorders;
4. The presence of clinically and/or hemodynamically significant congenital heart defects, defined as patients with congenital heart disease who already underwent or are awaiting surgical/percutaneous correction (including palliative cardiac surgery as Glenn and/or Fontan) or who are under current treatment with cardiac medications.
5. The presence of a hypersensibility known about sulpha drugs;
6. The presence of contraindications relative to the treatment by Bumetanide;
7. Patients already treated by diuretics;
8. Any of the following abnormal laboratory values at screening:

   * Hemoglobin <10 g/dL
   * Abnormal liver function defined as any 2 or more of the following: ≥3 × upper limit of normal (ULN) aspartate aminotransferase (AST), ≥3 × ULN alanine aminotransferase (ALT), ≥3 × ULN gamma-glutamyl transpeptidase (GGT), ≥3 × ULN alkaline phosphatase (ALP), or ≥2 × ULN total bilirubin
   * Abnormal liver function defined as any increase of ≥5 × ULN AST or ALT
   * Estimated glomerular filtration rate ≤80 mL/min/1.73 m2 (calculated by the Schwartz equation)
   * Plasma HCO3 > 32 i) A 12-lead ECG demonstrating QTc >450 msec at screening; j) Subject's weight less than 25 Kg.

k) Pregnancy as assessed by urine beta HCG

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual-Object long-term memory measures | Change from baseline (day 1) to 3 month (day 90 ± 3), day 150 ± 4
  Visual-Object Learning test (PROMEA, Vicari, 2007) - Efficacy criterion. Test assesses long-term visual memory skills.The total raw score of the visual episodic memory trial, the raw learning scores for each immediate recall trial (R_Score T1, T2, T3) and the raw score of the deferred recall trial (R_ Score Deferred) will be evaluated.

SECONDARY OUTCOMES:
Verbal long-term memory measure | Change from baseline (day 1) to 3 month (day 90 ± 3), day 150 ± 4
  Verbal Learning test (PROMEA, Vicari, 2007) - Efficacy criterion. Test assesses long-term verbal memory skills. The raw learning scores for each immediate recall trial (R_ScoreT1, T2, T3) and the raw score of the deferred recall trial (R_ Score Deferred) will be taken into account.
Visual-Spatial long-term memory measure | Change from baseline (day 1) to 3 month (day 90 ± 3), day 150 ± 4
  Visual-Spatial learning test (PROMEA, Vicari, 2007) - Efficacy criterion. Test assesses long-term spatial memory skills.The raw learning scores for each immediate recall trial (R_ScoreT1, T2, T3) and the raw score of the deferred recall trial (R_ Score Deferred) will be taken into account.
Long-term memory measures : recollection and familiarity | Change from baseline (day 1) to 3 month (day 90 ± 3), day 150 ± 4
  Processing Dissociation Procedure - PDP (Costanzo et al., 2013 - Efficacy criterion. Test assesses recollection and familiarity processes to memory performance..In the Processing Dissociation Procedures (PDP) test, of hits alarms responses (H) and false alarms responses (F) will be considered for both the "Inclusion" and "Exclusion" conditions.
Long-term memory measure: associative memory | Change from baseline (day 1) to 3 month (day 90 ± 3), day 150 ± 4
  Associative Memory (Costanzo et al., 2013) - Efficacy criterion. Test assesses recollection and familiarity processes to memory performance.The total raw scores for the "single item" and "associative item" condition and the learning raw scores for each trial of each condition (T1, T2, T3) will be evaluated.
Long-term measure - child's everyday memory | Change from baseline (day 1) to 3 month (day 90 ± 3), day 150 ± 4
  The Observer Memory Questionnaire-Parent Form (OMQ-PF, Gonzalez et al., 2008) - Likert scale questionnaire, test assesses parental beliefs about their child's everyday memory.For the assessment of everyday memory skills, the raw total score will be considered.
Adaptive level | Change from baseline (day 1) to 3 month (day 90 ± 3), day 150 ± 4
  ABAS II (Adaptive Behavior Assessment System Second Edition, Italian adaptation of Ferri R., Orsini A. e Rea M., Eds., 2014) - Efficacy criterion. Scale to obtain the parent's observations about the youth's behaviour and gives a complete overview of child and adolescent adaptive behaviours.
Executive measure | Change from baseline (day 1) to 3 month (day 90 ± 3), day 150 ± 4
  Behavior Rating Inventory Executive Function Second Edition (BRIEF 2, Gioia et al., 2000) Inventory evaluates everyday behaviors associated with EF in home and educational environments.The standardized scores (T) of Inhibit, Self-Monitor, Shift, Emotional Control, Initiate, Working Memory, Plan/Organize, Task-Monitor,and Organization of Materials scales will be evaluated. Behavioral Regulation Index (BRI), Emotional Regulation Index (ERI), Cognitive Regulation Index (CRI) and Global Executive Composite Score (GEC) also will be assessed.
Psychopathological measure - semi-structured diagnostic interview | Change from baseline (day 1) to 3 month (day 90 ± 3), day 150 ± 4
  K-Sads-Present and Lifetime Version (K-SADS-PL) (Kaufman et al., 2004) - Efficacy criterion. Interview assesses psychopathology according to the DSM-5 criteria.The total raw score related to current symptoms reported by the participant's parents in the interview and the symptom/disease decoding scores related to each diagnostic category will be evaluated.
Psychopathological measure - behavioral and psychopathological aspects | Change from baseline (day 1) to 3 month (day 90 ± 3), day 150 ± 4
  Conners' Parent Rating Scale -. Revised, Long Form (CPRS-R:L - Conners, 1997; Nobile, Alberti, & Zuddas, 2007) - Efficacy criterion. Questionnaire used parent's observations about the youth's behaviour and gives a complete overview of child and adolescent psychopathological disorders.The T scores of each scale of the questionnaire will also be evaluated.
Psychopathological measure - quantitative scale on anxiety symptoms | Change from baseline (day 1) to 3 month (day 90 ± 3), day 150 ± 4
  Multidimensional Anxiety Scale For Children - (MASC-parent report form March, 1997) - Efficacy criterion. Questionnaire assesses anxiety symptoms.The standardized total score (T) and T scores of the separation anxiety (SP), GAD, social anxiety (SAT), obsessions and compulsions (OC), physical symptoms (PS:T) and harm avoidance (HA) scales will be evaluated.
Psychopathological measure - behavioural and emotional problems | Change from baseline (day 1) to 3 month (day 90 ± 3), day 150 ± 4
  Child Behavior Checklist for Ages 6-18 - CBCL/6-18 (Achenbach e Rescorla, 2001) - Efficacy criterion. Questionnaire assesses behavioural and emotional problems in children and young people aged 6-18 years.The T-scores of each scale of the CBCL 6-18 questionnaire will be evaluated.
Quality of life | day 1/ day 7± 1/ day 31± 3/day 90 ± 3/day, day 150 ± 4
  PedsQL (PedsQL, JWVarni, 2004): measuring health-related quality of life (HRQOL) in healthy children and adolescents and those with acute and chronic health conditions. the raw scores of each scale (Physical , Emotional , Social , School) and the respective mean scores (Physical SC, Emotional Functioning ,Social Functioning , School Functioning), the physical index (T_Physical) , the psychosocial index (T_Psychosocial) and the mean total score (Total Score) of the questionnaire, will be evaluated.
Quality of sleep | day 1/ day 7± 1/ day 31± 3/day 90 ± 3/day, day 150 ± 4
  Sleep Disorders SDSC (The Sleep Disturbance Scale for Children, Bruni et al., 1996) - Sleepiness inventory is used to obtain the parent's observations about sleep disorders in children in five subdomains.T scores of each scale will be evaluated.
Bristol stool scale | Day 1, Day 7± 1, Day 31± 3, Day 90 ± 3, Day 150 ± 4
  Quality of life Stooling (based on Bristol stool scale) - Diagnostic medical tool designed to classify the form of human faeces into seven categories (Type 1-7)

OTHER OUTCOMES:
Biosample PBMC (blood) for biomarkers | Day 1 and Day 90 ±3
  Exploratory end-point - PBMCs will be analyzed from blood samples of all patients to identify possible biomarkers for response to treatment by evaluating the expression of NKCC1 and other genes (at RNA or protein levels)
Transcriptomic analysis by RNA-Seq assessment (on PBMCs samples) | Day 1, Day 90 ±3 and Day 150 ±4
  Exploratory end-point - All cohort patients will be analyzed for transcriptomic analysis by RNA-Seq. Total mRNA will be purified from PBMC and used for the mRNA-Seq library preparation
Genomic assessment (on blood samples) | Day 1
  Exploratory end-point - All participants will be analyzed by whole genome sequencing (both patients who respond to therapy and those who do not show any positive response). Genomic analysis will be performed on the pellet derived from centrifugation of the blood samples collected at visit 1, to obtain the corresponding plasma samples to be used for the proteomic analysis.
Proteomic (on plasma and PBMCs samples) assessment | Day 1, Day 90 ± 3 and Day 150 ± 4
  Exploratory end-point. Plasma and PBMC samples will be collected from all patients (both patients who respond to therapy and those who do not show any positive response). Five mL of peripheral venous blood samples x (supernatant) will be collected.
Metabolomic (on urine samples) assessment | Day 1, Day 90 ± 3 and Day 150 ± 4
  Exploratory end-point: Urine samples will be collected from all patients (both patients who respond to therapy and those who do not show any positive response) to identify possible biomarkers for treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Vicari, Principal Investigator — Bambino Gesù Children's Hospital
Locations (1):
- Bambino Gesù Children's Hospital, Rome, Italy

REFERENCES:
- [Background] Cancedda L, Fiumelli H, Chen K, Poo MM. Excitatory GABA action is essential for morphological maturation of cortical neurons in vivo. J Neurosci. 2007 May 9;27(19):5224-35. doi: 10.1523/JNEUROSCI.5169-06.2007. PMID 17494709
- [Background] Deidda G, Bozarth IF, Cancedda L. Modulation of GABAergic transmission in development and neurodevelopmental disorders: investigating physiology and pathology to gain therapeutic perspectives. Front Cell Neurosci. 2014 May 22;8:119. doi: 10.3389/fncel.2014.00119. eCollection 2014. PMID 24904277
- [Background] Savardi A, Borgogno M, De Vivo M, Cancedda L. Pharmacological tools to target NKCC1 in brain disorders. Trends Pharmacol Sci. 2021 Dec;42(12):1009-1034. doi: 10.1016/j.tips.2021.09.005. Epub 2021 Oct 4. PMID 34620512
- [Background] Lemonnier E, Degrez C, Phelep M, Tyzio R, Josse F, Grandgeorge M, Hadjikhani N, Ben-Ari Y. A randomised controlled trial of bumetanide in the treatment of autism in children. Transl Psychiatry. 2012 Dec 11;2(12):e202. doi: 10.1038/tp.2012.124. PMID 23233021
- [Background] Lemonnier E, Villeneuve N, Sonie S, Serret S, Rosier A, Roue M, Brosset P, Viellard M, Bernoux D, Rondeau S, Thummler S, Ravel D, Ben-Ari Y. Effects of bumetanide on neurobehavioral function in children and adolescents with autism spectrum disorders. Transl Psychiatry. 2017 May 9;7(5):e1124. doi: 10.1038/tp.2017.101. No abstract available. PMID 28485727